CLINICAL TRIAL: NCT05441592
Title: A Randomized Control Trial Assessing the Effect of Topical Tranexamic Acid on Risk of Hematoma in Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Edwin G. Wilkins, Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00210979
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Hematoma Postoperative
Keywords: Breast reduction; Gender-affirming mastectomy; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Irrigation that contains tranexamic acid (TXA) (Experimental)
  Interventions: Drug: Tranexamic acid injection
- No additional irrigation usual care (Other)
  Interventions: Other: No additional irrigation

INTERVENTIONS:
Drug: Tranexamic acid injection — The breast pockets will additionally be irrigated with 150 cc of 2.67% TXA (75 cc in each breast). The TXA solution will be allowed to be sit in the breast pocket for 15 minutes and then removed after 15 minutes.
  Arms: Irrigation that contains tranexamic acid (TXA)
Other: No additional irrigation — There will be no additional irrigation after the standard surgical procedure.
  Arms: No additional irrigation usual care

SUMMARY:
This trial is being completed to evaluate the safety and efficacy of topical tranexamic acid use in preventing hematomas in routine breast plastic surgery operations.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral breast reduction or bilateral gender-affirming mastectomy
* For patients undergoing bilateral breast reduction, any skin incision pattern or pedicle is acceptable.
* For patients undergoing bilateral gender-affirming mastectomy, any skin incision and mastectomy type is acceptable

Exclusion Criteria:

* Active thromboembolic disease or history of intrinsic risk of thrombosis or thromboembolism, including retinal vein or artery occlusion
* Current use of systemic anticoagulation
* Hypersensitivity to tranexamic acid
* Concomitant use of combined hormonal contraceptives
* Use of factor IX complex concentrates, anti-inhibitor coagulant concentrates or all-trans retinoic acid
* History of acquired defective color vision
* History of subarachnoid hemorrhage
* Pregnancy
* History of renal impairment or serum Creatinine >1.5 milligrams per deciliter (mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Wilkins, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Irrigation that contains tranexamic acid (TXA) | No additional irrigation usual care
Started | 55 | 52
Completed | 54 | 47
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irrigation That Contains Tranexamic Acid (TXA) | No Additional Irrigation Usual Care | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 31] | 28 [22 to 33] | 26 [21 to 32]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 0 | 0 | 0
  Transgender Female | 0 | 0 | 0
  Transgender Male | 34 | 25 | 59
  Non-Binary | 14 | 11 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 43 | 41 | 84
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 55 | 52 | 107

OUTCOME MEASURES:

1. Primary Outcome: Hematomas
Description: Results reflect the number of hematomas that occurred during the trial, requiring operative washout or aspiration in participants who received TXA versus participants who did not receive TXA.
Time Frame: Up to approximately 4 weeks after surgery
Measure: Number; unit: hematomas
Arm/Group | Irrigation that contains tranexamic acid (TXA) | No additional irrigation usual care
Number analyzed (Participants) | 54 | 47
hematomas | 0 | 1
Statistical Analysis 1: Comparison: Irrigation that contains tranexamic acid (TXA) vs No additional irrigation usual care; Test type: Superiority; p = 0.486, Fisher Exact

2. Secondary Outcome: Participants Who Experienced a Major Thromboembolic Event Related to the Study Drug
Description: Results reflect the number of participants who experienced any major thromboembolic event during the trial. Major thromboembolic events included, but were not limited to, deep vein thrombosis, pulmonary embolism, and stroke.
Time Frame: Up to approximately 4 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Irrigation that contains tranexamic acid (TXA) | No additional irrigation usual care
Number analyzed (Participants) | 54 | 47
Participants | 0 | 0

3. Secondary Outcome: Participants Who Experienced Major Complications Other Than Hematoma
Description: Results reflect the number of participants who experienced any major complication other than a hematoma. Major complications included, but were not limited to, infection, seroma, hypersensitivity reaction to TXA, and renal impairment.
Time Frame: Up to approximately 4 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Irrigation that contains tranexamic acid (TXA) | No additional irrigation usual care
Number analyzed (Participants) | 54 | 47
Participants | 0 | 2
Statistical Analysis 1: Comparison: Irrigation that contains tranexamic acid (TXA) vs No additional irrigation usual care; Test type: Superiority; p = 0.234, Fisher Exact

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Irrigation that contains tranexamic acid (TXA) | No additional irrigation usual care
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/55 | 1/52
Other Adverse Events (participants affected / at risk) | 6/55 | 6/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irrigation that contains tranexamic acid (TXA) (N=55) | No additional irrigation usual care (N=52)
Hematoma Requiring Reoperation (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irrigation that contains tranexamic acid (TXA) (N=55) | No additional irrigation usual care (N=52)
Surgical site infection (Infections and infestations) | 0 | 2
Delayed wound healing (Injury, poisoning and procedural complications) | 4 | 5
Rash/Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT05441592/Prot_SAP_000.pdf